CLINICAL TRIAL: NCT01778725
Title: S100B as a Marker for Fetal Brain Injury in Premature Rupture of Membranes
Brief Title: Early Identification of Brain Insult in Chorioamnionitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-12-9616-BW-CTIL
Record Dates: First submitted 2012-11-25; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Chorioamnionitis; Cerebral Palsy
Keywords: Chorioamnionitis, S100B, Brain, Neuro-development
MeSH Terms: conditions — Chorioamnionitis; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Premature breaking of the amniotic fluids during pregnancy caries high risk for infection of the amniotic fluid. One of the results of chorioamnionitis is brain injury of the fetus. Fetus' brain is highly vulnerable and could be harmed even by mild inflammation before fulminant infection is developed. The aim of this study is to identify, as early as, possible signs of brain injury. S100B protein will be used as a marker for brain insult. S100b level were associated with the occurrence and size of stroke and brain trauma in adults and children. Moreover, S100B crosses the membrane and its level in women with preterm labor was associated with brain injury of preterm infant.

The study question is whether the levels of S100B in women with early amniotic fluids breakdown are associated with future brain injury of the infant, as assessed by head ultrasound and neurological examination.

ELIGIBILITY:
Inclusion Criteria:

* Rupture of the amniotic sac before 32 weeks
* Gestational age less than 32 weeks
* Singleton

Exclusion Criteria:

* Intrauterine growth restriction
* Positive TORCH
* Fetus' brain malformation
* Fetus' brain hemorrhage
* Maternal medication with teratogenic effect

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with premature rupture of the amniotic sac.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Developmental assessment | 18 month
  Developmental assessment at 18 month
  1. Vineland Adaptive Behavior Scales
  2. Griffith Mental Development Scales
Developmental assessment | 3 month
  Developmental assessment at term and 3 month
  1. Neurological examination
  2. Test of infant motor performance

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Weisz, M.D., Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Seba Medical Center, Ramat Gan, Israel